CLINICAL TRIAL: NCT02835976
Title: A Single-Center, Open-Label, Single Oral Dose Phase I Study to Determine the Excretion Balance of Radiocarbon (i.e., the Sum of 14C-Labeled TRO19622 and Its 14C-Metabolites) and to Investigate the Pharmacokinetics and Metabolic Profile of TRO19622
Brief Title: A Study of the Excretion Balance of Radiocarbon and the Pharmacokinetics and Metabolic Profile of TRO19622 (Olesoxime)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trophos SA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP29867; 2014-002470-37 (EudraCT Number)
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — olesoxime

ARMS (1):
- Olesoxime (Experimental): Participants will receive a single dose of liquid suspension of 14C-labeled olesoxime containing an equivalent of 600 milligrams (mg) of the compound. The total amount of administered radiocarbon will be 93 microcuries (mcCi), or 3.447 megabecquerels (MBq).
  Interventions: Drug: Olesoxime

INTERVENTIONS:
Drug: Olesoxime — Olesoxime will be given orally on Day 1 as a 600-mg liquid suspension within 30 minutes after starting a standardized high-fat breakfast.
  Other Names: TRO19622

SUMMARY:
This Phase I study is designed to determine the excretion balance of radiocarbon, as the sum of carbon-14 (14C)-labeled TRO19622 and its 14C-metabolites, and to investigate the pharmacokinetics and metabolic profile of TRO19622 (olesoxime) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 20.0 to 28.0 kilograms per meter-squared (kg/m^2) and body weight at least 60 kilograms (kg)
* Fitzpatrick skin type less than (<) 4
* Good health according to medical history, physical examination, laboratory parameters, vital signs, and 12-lead electrocardiogram (ECG)
* Negative urine test for drugs of abuse
* Negative alcohol breath test
* Negative tests for hepatitis or human immunodeficiency virus (HIV)
* Use of effective contraception during and for 3 months beyond study participant, among sexually active non-vasectomized participants with females partners of childbearing potential

Exclusion Criteria:

* Concomitant or recent medication use within 2 weeks prior to Day 1, except for paracetamol
* Use of enzyme-inducing drugs within 2 months prior to Day 1
* Any medical condition that may alter the pharmacokinetics of olesoxime or affect interpretation of study results
* Irregular bowel movements
* Drug addiction or alcoholism
* Use of nicotine products
* Participation in another clinical study within 12 weeks prior to Day 1
* Exposure to ionizing radiation within one year prior to Day 1

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
T1/2 of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Apparent Plasma Clearance (CL/F) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
CL/F of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Apparent Volume of Distribution (Vz/F) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
Vz/F of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Cumulative Amount of Olesoxime Excreted in Urine | Continuous urine collection from pre-dose (0 h) to post-dose (432 h, or until release criteria are met) following single dose on Day 1
Cumulative Amount of Olesoxime Excreted in Expired Air | Pre-dose (0 h) and post-dose (8, 10, 12, 16, 24, 48, 72, 96 h) following single dose on Day 1
Cumulative Amount of Olesoxime Excreted in Feces | Continuous fecal collection from pre-dose (0 h) to post-dose (432 h, or until release criteria are met) following single dose on Day 1
Renal Clearance (CLr) of Olesoxime | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
AUClast of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
AUCinf of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Percentage of Participants with Adverse Events (AEs) | Continuously from Screening until 7 days after last dose (up to 46 days overall)
Maximum Observed Concentration (Cmax) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 hours [h]) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
Cmax of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Time of Maximum Observed Concentration (Tmax) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
Tmax of Radiocarbon | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 168, 216, 264, 312, 360, 408 h) following single dose on Day 1
Area Under the Concentration-Time Curve from Drug Administration to Last Quantifiable Concentration (AUClast) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUCinf) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1
Elimination Half-Life (t1/2) of Olesoxime and Any Major Metabolite(s) Identified | Pre-dose (0 h) and post-dose (2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408 h) following single dose on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche